CLINICAL TRIAL: NCT04653155
Title: Cognitive Behavioural Therapy for Insomnia for Chinese Adults: a Randomized Controlled Trial
Brief Title: Cognitive Behavioural Therapy for Insomnia for Chinese Adults: a RCT
Acronym: CBTI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Kwok Pui Ling Amy, Clinical Psychologist, Hospital Authority, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2019.126
Record Dates: First submitted 2020-08-14; First posted 2020-12-04 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Insomnia
Keywords: Cognitive behaviour therapy, group treatment, insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Participants in the treatment group will show significant improvement on insomnia symptoms after intervention compared to those in the waitlist control group.
  Interventions: Behavioral: Cognitive behavioural therapy for insomnia
- Waitlist control (No Intervention): Participants in the waitlist control group will show little improvement on insomnia symptoms after the treatment period of the treatment group.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy for insomnia — Cognitive behavioural therapy for insomnia
  Arms: Treatment arm

SUMMARY:
Background: Insomnia is a common mental problem, where people experienced difficulty falling asleep, problem maintaining asleep and early morning awakening. It is highly prevalent world-wide and in Hong Kong, causing significant suffering and distress. While evidence based intervention exists, e.g. cognitive-behavioural therapy (CBT), there will not enough therapists to meet treatment demand. A more efficient delivery of treatment, e.g. internet based therapy is called for that can delivery treatment more cost efficiently by requiring lesser therapist time.

Objective: This study aims at evaluating the effectiveness of CBTi (Gp) on treating Chinese insomniac adults in Hong Kong. There has been criticism that most clinical trials have been conducted with Caucasians in Western countries and little has been done with ethnic minorities, including Asians in these countries, not to mention Asians in Asian countries, e.g., Chinese in Hong Kong.

Design: A two-arm parallel-group randomised controlled trial, comparing the treatment and waitlist group

Method: A CBTi protocol would be developed. Approximately 60 Chinese adults with insomnia will be recruited in Hong Kong and randomised into one of the two groups (treatment vs. waitlist). The treatment last for 6 weeks, plus a 3-month follow-up period. The primary outcome measure will be Insomnia Severity Index (ISI).

DETAILED DESCRIPTION:
Insomnia is characterized by difficulty in initiating sleep, difficulty in maintaining sleep, early morning awakening and non-restorative sleep, which should be relatively frequent (>/= 3 times/ week), persistent (>/= 2-4 weeks) and severe enough to affect daytime functioning. It is among the most common mental disorders. Epidemiological surveys in Western countries found a high prevalence of insomnia syndrome (9.2-13%) and insomnia symptoms (11.4% to 38%). In Hong Kong, a prevalence of 11.9% was reported for community adults. Given such high prevalence, insomnia is evidently one major health concern across diverse communities, including Hong Kong. Furthermore, the disorder runs a chronic and debilitating course if untreated.

Interrelationships between insomnia and mental health are now well established in the epidemiological literature, with insomnia shown to be frequently comorbid with mental health concerns, such as depression or anxiety and risk of suicide. Insomnia symptoms have repeatedly been shown to increase the risk of subsequent depression. Also, it is shown that augmenting an antidepressant medication with a brief, symptom focused, cognitive-behavioral therapy for insomnia is promising for individuals with depression and comorbid insomnia in terms of alleviating both depression and insomnia. It is clear that insomnia is not only a disorder of high personal suffering, but is also associated with high and recurring societal costs. These facts strongly argue for the need of effective treatments to relieve personal suffering, caring burdens, and societal economic costs.

Fortunately, there are effective treatments available for insomnia, particularly cognitive-behavioural therapy (CBT). In a number of meta-analysis of insomnia treatments, CBT is effective and consistently performs better than placebo and other control conditions in improving nighttime insomnia symptoms, including sleep latency, total sleep time, wake after sleep onset, and insomnia symptoms. CBT for insomnia (CBTi) packages include stimulus control, relaxation, sleep restriction and their combination meet APA criteria for empirically validated treatment for insomnia based on the strength of results from a number of empirical studies.

Unfortunately, while effective psychological treatments exist, there is only limited manpower to provide the intervention. Western studies showed that 15-25% of children and adults were suffering from mental health disorders, but only 20-30% of them had access to treatment. Locally in Hong Kong, we are facing an almost identical situation. About 15% of children and adults suffered from mental health disorders, but again only 15-30% of them had access to mental health services. Obviously, a shortage of mental health professionals such as psychiatrists or clinical psychologists is a worldwide phenomenon. In Hong Kong, our situation regarding the availability of clinical psychologists (CPs) in providing psychological treatment is even worse. We have a ratio of approximately 1 CP to 18,000 in the Hong Kong population, far below the ratio of 1 in 3,500 in the USA.

Most governments, including those of richer countries like USA, will admit that they will never have the resources to increase the number of mental health professionals like psychiatrists and CPs to meet the societal demand. Instead, a more viable solution is to look for greater cost-efficiency in delivering services. Recent meta-analyses find the effectiveness of group psychological treatment (mostly CBT) for insomnia as largely comparable to that of traditional one on one therapy. Group therapy is thus advocated as a less-intensive, cost-effective way to offer evidence-based treatment.

Based on Morin, we developed a treatment protocol for CBTi, incorporating both education and individualized feedback. The protocol implements all of the key procedures in one-on-one CBTi such as sleep restriction, stimulus control, managing dysfunctional beliefs about sleep, behavioural experiments, increasing energizing behaviours, all of which target the maintaining factors of insomnia. Patients would be assigned a therapist to follow up on them via either brief (5-10 minutes) telephone calls. Compared to traditional face to face CBTi, the protocol requires 32% of the therapist's time of the latter, i.e., a 68% drop in the therapist's time.

There is a paucity of study in the effectiveness of cognitive behaviour therapy for insomnia in Hong Kong Chinese, let alone CBTi in group. This proposal aims at developing a CBTi protocol for treatment of insomnia in Hong Kong to increase the access of evidence-based treatment to local Chinese insomnia adults. This involves protocol development, test-run and a randomized controlled trial (RCT) with a waitlist control group and a short-term follow-up of three months.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia
* Chinese aged 18-65 years old
* Chinese reading and writing proficiency of primary school
* Ability to give consent
* Accept randomization

Exclusion Criteria:

* substance abuse or dependence
* manic or hypomanic episode
* schizophrenia
* personality disorders
* posttraumatic stress disorder (PTSD)
* mental retardation
* organic mental disorder
* Suicidal risk or a suicidal attempt in the past three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Insomnia Symptom Inventory (ISI) (Bastien et al, 2001) | Change from baseline Insomnia Symptom Inventory at 3 months
  A 7-item self-report questionnaire assessing the nature, severity and the impact of insomnia. Insomnia Symptom Inventory is the primary outcome measure. All items are assessed on a 5-point scale (0-4), with its total score ranging between 0 to 28. Higher score representing worse insomnia symptoms.

SECONDARY OUTCOMES:
Change in Dysfunctional Beliefs about Sleep Scale (DBAS) (Morin et al, 2007) | Change from baseline Dysfunctional Beliefs about Sleep Scale at 3 months
  A self-report questionnaire for evaluation of cognition, behaviours and attitudes related to insomnia. All items are assessed on a 5-point scale (0-4). Its total score ranged between 0 to 112, with higher score representing more dysfunctional beliefs about sleep.
Change in Patient Health Questionnaire 9 (PHQ-9) (Kroenke & Spitzer, 2002) | Change from baseline Patient Health Questionnaire 9 (PHQ-9) at 3 months
  A 9-item self-report questionnaires for evaluation of depression. All items are assessed on a 4-point scale (0-3). Its total score ranged between 0 to 27, with higher score representing more severe depressive symptoms.
Change in Generalized Anxiety Disorder-7 item (GAD-7) Questionnaire (Spitzer et al, 2006) | Change from baseline Generalized Anxiety Disorder-7 item (GAD-7) Questionnaire at 3 months
  A 7-item self-report questionnaires for evaluation of general anxiety. All items are assessed on a 4-point scale (0-3), with its total score ranging between 0 to 21. Higher score representing increased anxiety symptoms.
Change in Work and Social Adjustment Scale (WSAS) (Mundt et al, 2002) | Change from baseline Work and Social Adjustment Scale at 3 months
  A 5-item simple self-report measure of impairment in functioning. All items are assessed on a 9-point scale (0-8), with its total score ranging between 0 to 40. Higher score representing greater impairment in functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Psychology, New Territories East Cluster, Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No